CLINICAL TRIAL: NCT00455767
Title: Phase IIA Multicenter 1 Week Treatment, Randomised, Double-Blind, Placebo Controlled Study of Depelestat in Patients Suffering From Acute Respiratory Distress Syndrome
Brief Title: Safety and Efficacy Study of Depelestat in Acute Respiratory Distress Syndrome (ARDS) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: François Saudubray, M.D., Debiopharm S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEB-EPIV-201; 2006-000756-41 (EUDRACT NR)
Record Dates: First submitted 2007-03-14; First posted 2007-04-04 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Fibrosis; Lung Disease; Respiratory Disorders; Respiratory Distress Syndrome, Adult; Acute Respiratory Distress Syndrome; Pulmonary Fibrosis; Inflammation
Keywords: persistent ARDS; alveolar inflammation; early pulmonary fibrosis; mechanichal ventilation; P/V curve; Static compliance; elastase activity; inhibitor of Human Neutrophil Elastase
MeSH Terms: conditions — Fibrosis; Lung Diseases; Respiration Disorders; Respiratory Distress Syndrome; Pulmonary Fibrosis; Inflammation | interventions — depelestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Depelestat
  Interventions: Drug: EPI-hNE4
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EPI-hNE4 — I.V. injection of 1mg/kg Depelestat (EPI-hNE4) 3 times daily for 7 days
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The study is aimed to assess safety of Depelestat treatment, as well as efficacy on prevention and treatment of alveolar inflammation in early pulmonary fibrosis in patients suffering from persistent Acute Respiratory Distress Syndrome.

DETAILED DESCRIPTION:
This is a multicenter, randomised, double-blind, parallel groups, placebo-controlled, 1 week treatment of Depelestat, in patients suffering from persistent ARDS.

Patients admitted in the intensive care unit presenting ARDS criteria persistent for 12 hours to 24 hours, will be randomly assigned to the treatment by Depelestat or placebo, after a pre-treatment period as short as possible with a maximum of 48 hours since ARDS criteria are met. During the pre-treatment period, the informed consent will be obtained from the legally authorized relative of the patient, and pre-treatment biological and functional examinations will be performed, particularly blood samples and BAL for biological parameters measurement, and ventilatory mechanics, for assessment of static compliance of the respiratory system.

After the pre-treatment period, the patient will receive treatment by Depelestat or placebo during 7 days, or until extubation of the patient if this occurs before 7 days of treatment. During this treatment period, the patient will be submitted to a daily measurement of static compliance of the respiratory system, as long as the patient adaptation to 24 hours after mechanical ventilation allows the procedure, and at 96 initiation of treatment, to a blood sampling and a bronchoalveolar lavage for several biological parameters assessment.

On the first and last day of administration, blood will be also collected for pharmacokinetic evaluation.

During the post-treatment period, the patient will be submitted, at 48 h ± 24 h after the end of treatment, to a blood sampling and a BAL (this BAL is not performed when contraindication criteria are present, if the patient is already extubated, and in case of planed extubation during the subsequent 24 hours) for several biological parameters assessment, and a daily measurement of static compliance as long as the patient adaptation to mechanical ventilation allows the procedure. Patients already extubated will not be submitted to BAL nor to static compliance measurements.

After the end of the treatment, patients will be followed daily for 28 days after the diagnostic of ARDS, or until death whichever occurred first.

The duration of the study for each survivor patient will be 28 days. Survivors to day 28 will be contacted monthly to assess survival and fill in a QOL questionnaire on days 60 and 90.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from persistent ARDS as defined by the American and European Consensus Conference on ARDS, 1994

Exclusion Criteria:

* ARDS secondary to traumatism
* Pulmonary emphysema on pulmonary fibrosis
* Lung pneumocystosis
* Bronchopleural fistula
* Systemic corticosteroid treatment for more than 2 weeks before inclusion
* Severe organ disease excepted renal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Static compliance relative change from pre-treatment to last on treatment

SECONDARY OUTCOMES:
PCPIII and cytokines concentration, as well as neutrophil influx relative change in BAL fluid from pre-treatment to post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: François Saudubray, MD, Study Director — Debiopharm SA
Locations (14):
- France (11):
  - Alain Mercat, Angers
  - Yves Castaing, Bordeaux
  - Laurent Brochard, Créteil
  - Jean-François Timsit, Grenoble
  - Claude Guerin, Lyon
  - Samir Jaber, Montpellier
  - Jean-Jacques Rouby, Paris
  - Jean-Daniel Chiche, Paris
  - Jean-Yves Fagon, Paris
  - Jean-Christophe Richard, Rouen
  - Jean-Michel Arnal, Toulon
- Massimo Antonelli, Roma, Italy
- Jordi Mancebo D., Barcelona, Spain
- Fekri Abroug, Monastir, Tunisia

REFERENCES:
- [Background] Honore S, Attalah HL, Azoulay E, Soussy CJ, Saudubray F, Harf A, Brochard L, Delclaux C. Beneficial effect of an inhibitor of leukocyte elastase (EPI-hNE-4) in presence of repeated lung injuries. Shock. 2004 Aug;22(2):131-6. doi: 10.1097/01.shk.0000126861.77543.d0. PMID 15257085
- See also: Related Info — http://www.ncbi.nlm.nih.gov/